CLINICAL TRIAL: NCT06448247
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of SPY001-001 in Healthy Participants
Brief Title: A Study of SPY001-001 in Healthy Volunteers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Spyre Therapeutics, Inc. (Industry)
Collaborators: Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SPY001-101
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- SAD Cohorts 1-5 Experimental Arm (Experimental): Participants will receive a single dose of SPY001-001 in a dose escalation format
  Interventions: Drug: SPY001-001
- SAD Cohorts 1-5 Placebo Arm (Placebo Comparator): Participants will receive a single dose of placebo
  Interventions: Other: Placebo
- MAD Cohorts 1-3 Experimental Arm (Experimental): Participants will receive two doses of SPY001-001 in a dose escalation format
  Interventions: Drug: SPY001-001
- MAD Cohorts 1-3 Placebo Arm (Placebo Comparator): Participants will receive two doses of placebo
  Interventions: Other: Placebo
- SAD Cohorts 6-7 Experimental Arm (Experimental): Participants of Japanese descent will receive a single dose of SPY001-001
  Interventions: Drug: SPY001-001
- SAD Cohorts 6-7 Placebo Arm (Placebo Comparator): Participants of Japanese descent will receive a single dose of placebo
  Interventions: Other: Placebo
- SAD Cohorts 8-9 Experimental Arm (Experimental): Participants of Chinese descent will receive a single dose of SPY001-001
  Interventions: Drug: SPY001-001
- SAD Cohorts 8-9 Placebo Arm (Placebo Comparator): Participants of Chinese descent will receive a single dose of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SPY001-001 — Experimental
  Arms: MAD Cohorts 1-3 Experimental Arm; SAD Cohorts 1-5 Experimental Arm; SAD Cohorts 6-7 Experimental Arm; SAD Cohorts 8-9 Experimental Arm
Other: Placebo — Placebo
  Arms: MAD Cohorts 1-3 Placebo Arm; SAD Cohorts 1-5 Placebo Arm; SAD Cohorts 6-7 Placebo Arm; SAD Cohorts 8-9 Placebo Arm

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single- and multiple-dose, first in human safety, tolerability, and pharmacokinetic study of SPY001-001 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Willing and able to attend the necessary visits to the CRU, comply with all testing requirements, remain at the study site unit for the duration of the confinement period and return for the outpatient visits

Exclusion Criteria:

* Participation in more than one cohort
* Evidence of clinically significant abnormality or disease
* Known history of illicit drug use or drug abuse, harmful alcohol use or alcoholism, and/or smoking or nicotine-containing product use within 3 months prior to the first dose of study drug
* History of severe allergic reactions or hypersensitivity
* Donation or loss of >1 unit of whole blood within 1 month prior to dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events | Up to 64 weeks
  Incidence, severity, and causal relationship of TEAEs

SECONDARY OUTCOMES:
Cmax | Up to 64 weeks
  Maximum concentration after single and multiple ascending doses
Tmax | Up to 64 weeks
  Time to reach maximum concentration after single and multiple ascending doses
t1/2 | Up to 64 weeks
  Half life after single and multiple doses
AUC | Up to 64 weeks
  Area under the curve after single and multiple ascending doses
ADA | Up to 64 weeks
  Incidence of anti-drug antibody after single and multiple ascending doses

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Nguyen, MD, Study Chair — Spyre Therapeutics
Locations (2):
- Spyre Site 2, Cypress, California, United States
- Spyre Site 1, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No